CLINICAL TRIAL: NCT00073892
Title: A Phase I/II Study Of PI-88 In Advanced Malignancies (Phase I), And In Advanced Melanoma(Phase II)
Brief Title: PI-88 in Treating Patients With an Advanced Malignancy (Cancer) or Stage IV Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellxpert Biotechnology Corp. (Industry)
Collaborators: Medigen Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROGEN-PR88201; CDR0000335412 (Registry Identifier: PDQ (Physician Data Query)); COMIRB-01-207
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Melanoma (Skin); Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — phosphomannopentaose sulfate

ARMS (1):
- PI-88 (Experimental): Patients receive four consecutive days treatment each week in a 4-week cycle.
  Interventions: Drug: PI-88

INTERVENTIONS:
Drug: PI-88 — 250 mg/day injected subcutaneously on four consecutive days each week in a 4- week cycle
  Other Names: Mannopentaose phosphate sulfate

SUMMARY:
RATIONALE: PI-88 may stop the growth of cancer by stopping blood flow to the tumor.

PURPOSE: Phase I/II trial to study the effectiveness of PI-88 in treating patients who have an advanced malignancy (cancer) or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Phase I

* Determine the maximum tolerated dose of PI-88 in patients with an advanced malignancy.
* Determine the safety and tolerability of this drug in these patients.

Phase II

* Determine the progression-free survival and time to progression in patients with stage IV melanoma treated with this drug.
* Determine the biological activity of this drug in these patients.

OUTLINE: This is an open-label, dose-escalation study.

* Phase I (parts 1 and 2):

  * Part 1: Patients receive PI-88 subcutaneously (SC) once daily on days 1-4 and 15-18.

Cohorts of 3-6 patients receive escalating doses of PI-88 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD has been determined in part I, the effect of dose frequency is determined in patients in part II.

* Part 2: Patients receive PI-88 SC once daily on days 1-4, 8-11, 15-18, and 22-25 at a dose based on the MTD determined in part 1.

Cohorts of 3 patients receive escalating doses of PI-88 until the MTD at this frequency is determined.

* Phase II (patients with metastatic melanoma): Patients receive PI-88 as in phase I, part 2 at the MTD.

Treatment in both phases repeats every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 18-69 patients (18-30 for phase I [part 1], 6-9 for phase I [part 2], and 25-30 for phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Phase I

* Histologically or cytologically confirmed malignancy
* No other effective treatment available OR failed prior therapy
* No prior or concurrent symptomatic or known CNS involvement or brain or meningeal metastases

Phase II

* Diagnosis of stage IV melanoma
* Metastatic disease must be measurable
* No other effective treatment available OR failed prior therapy
* Asymptomatic brain metastases allowed provided patient is off steroids

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 70-100%

Life expectancy

* At least 3 months

Hematopoietic

* Neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Negative serotonin release assay test for anti-heparin antibodies
* No other abnormal bleeding tendency
* No history of heparin-induced thrombocytopenia
* No history of immune-mediated thrombocytopenia
* No history of thrombolytic thrombocytopenic purpura
* No history of other platelet disease

Hepatic

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* AST and ALT no greater than 2 times ULN (5 times ULN if liver metastases are present)
* PTT normal (20-34 sec)
* PT less than 1.5 times ULN

Renal

* Creatinine clearance greater than 60 mL/min OR
* Glomerular filtration rate greater than 60 mL/min

Cardiovascular

* No myocardial infarction within the past 3 months
* No stroke within the past 3 months
* No congestive heart failure within the past 3 months

Gastrointestinal

* No history of acute or chronic gastrointestinal bleeding within the past 2 years
* No inflammatory bowel disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No AIDS-related illness
* No serious infection within the past 4 weeks
* No history of alcohol, drug, or other substance abuse
* No history of allergy and/or hypersensitivity to anti-coagulants/thrombolytic agents (e.g., heparin)
* No risk of bleeding due to open wounds or planned surgery
* No clinically significant nonmalignant disease
* No uncontrolled infection

Inclusion Criteria

* Current diagnosis of metastatic melanoma, where other effective therapy was not available or had failed.
* Measurable disease. Metastatic lesions had to have been measurable by MRI or CT, and cutaneous lesions by physical examination.
* Biopsiable Lesion Group only: Must have had at least one biopsiable lesion that was bi-dimensionally measurable and previously unirradiated.
* Age≥ 18 years.
* Have voluntarily given written informed consent to participate in this study.
* Performance status: ECOG 0 - 2 (Karnofsky 70 -100%).
* Life expectancy of at least 3 months.
* Neutrophil count > 1.5 x 109/L (1,500/mm3).
* Platelet count > 100 x 109/L (100,000/mm3).
* APTT normal (20 - 34 sec).
* PT <1.5 x ULN.
* Calculated creatinine clearance, using the Cockcroft-Gault formula, >60 mL/min. If just below 60 mL/min, then GFR>60 mL/min as determined by EDTA or DTPA scan.
* Bilirubin <1.5 x ULN.
* AST and ALT up to 2 x ULN; except in the presence of liver metastases; up to 5 x ULN.

Exclusion Criteria

* Current symptomatic central nervous system involvement, or active brain or meningeal metastases.
* Concomitant use of aspirin (> 100 mg/day), non-steroidal anti-inflammatory drugs (with the exception of COX-2 inhibitors), heparin, low molecular weight heparin or warfarin (> 1 mg/day) which was ongoing or anticipated during the study period. Low-dose aspirin (100 mg/day or less) or low-dose warfarin (1 mg/day or less) was permitted.
* Heparin or low molecular weight heparin within the previous 2 weeks.
* Chemotherapy, investigational therapy or hormonal therapy in the previous 4 weeks.
* Radiotherapy to a major bone marrow bearing area such as pelvis, femoral heads, lumbar-sacral spine, within the previous 4 weeks. Radiotherapy to other sites within the previous 2 weeks.
* History of allergy and/or hypersensitivity to anti-coagulants/thrombolytic agents, especially heparin.
* History of heparin-induced thrombocytopenia, immune mediated thrombocytopenia, thrombotic thrombocytopenic purpura and/or other platelet diseases, or laboratory evidence of anti-heparin antibodies.
* Myocardial infarction, stroke or congestive heart failure within the previous 3 months
* History of acute or chronic gastrointestinal bleeding within the previous two years, inflammatory bowel disease, any other abnormal bleeding tendency, or patients at risk of bleeding due to open wounds or planned surgery.
* Uncontrolled infection or serious infection within the previous 4 weeks.
* Clinically significant non-malignant disease.
* Known AIDS-related illness or HIV positive.
* Women who were pregnant, breast feeding, or of childbearing potential in whom pregnancy could not be excluded.
* History of abuse of alcohol, drugs or other substances.
* Not recovered from major surgery if conducted prior to the study.

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* More than 4 weeks since prior chemotherapy

Endocrine therapy

* More than 4 weeks since prior hormonal therapy

Radiotherapy

* More than 2 weeks since prior radiotherapy
* More than 4 weeks since prior radiotherapy to a major bone-marrow bearing area (e.g., pelvis, femoral heads, or lumbar-sacral spine)
* Concurrent palliative radiotherapy allowed

Surgery

* Recovered from prior major surgery
* No concurrent surgery

Other

* More than 2 weeks since prior heparin or low-molecular weight heparin
* More than 4 weeks since other prior investigational therapy
* No other concurrent investigational drugs
* No other concurrent antineoplastic therapy
* No concurrent aspirin or aspirin-containing medications
* No concurrent nonsteroidal anti-inflammatory drugs

  * Concurrent cyclooxygenase-2 inhibitors allowed
* No concurrent heparin or low-molecular weight heparin
* No concurrent warfarin or warfarin-containing medications
* No other concurrent anticoagulant medications

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-01; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Efficacy Analysis | end of Cycle 6 of study treatment (24 weeks)
  non-progression rate (objective response or stable disease)

SECONDARY OUTCOMES:
Efficacy Analysis | were time to progressive disease, survival, duration of partial response, complete response and stable disease
  time to progression and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: S. G. Eckhardt, MD, Principal Investigator — University of Colorado, Denver
Locations (5):
- University of Colorado Cancer Center at University of Colorado Health Sciences Center, Aurora, Colorado, United States
- Australia (4):
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Queen Elizabeth Hospital, Woodville, South Australia
  - Alfred Hospital, Melbourne, Victoria
  - Sir Charles Gairdner Hospital - Perth, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided